CLINICAL TRIAL: NCT06274554
Title: A Prospective, Randomized, Placebo-controlled Trial of Fluconazole in Combination With IL-23 Therapy Versus IL-23 Therapy Alone for the Treatment of Crohn's Disease
Brief Title: Testing the Role of Anti-fungal Therapy in Improving the Response to Therapies for Crohn's Disease
Acronym: FUN-CD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-11026746
Record Dates: First submitted 2024-02-15; First posted 2024-02-23 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Crohn's Disease; Inflammatory Bowel Diseases
Keywords: Fluconazole; IL-23
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Fluconazole; risankizumab; Ustekinumab; guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blinded study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IL-23 Therapy with Fluconazole (Experimental): Fluconazole will be blindly administered as capsules for oral consumption. On the first day, 200 mg will be given. Subjects will then take 100 mg once daily for thirteen days.
  Interventions: Drug: Fluconazole; Biological: IL-23 Therapy
- IL-23 Therapy with Placebo (Placebo Comparator): Placebo will be blindly administered as capsules for oral consumption. On the first day, 200 mg will be given. Subjects will then take 100 mg once daily for thirteen days.
  Interventions: Drug: Placebo; Biological: IL-23 Therapy

INTERVENTIONS:
Drug: Fluconazole — Oral fluconazole capsules.
  Other Names: Diflucan
  Arms: IL-23 Therapy with Fluconazole
Drug: Placebo — Oral placebo capsules will be used as a comparator.
  Arms: IL-23 Therapy with Placebo
Biological: IL-23 Therapy — Risankizumab (IL-23), Guselkumab (IL-23), or Ustekinumab (IL-12/23) as standard of care treatment.
  Other Names: Risankizumab; Ustekinumab; Guselkumab

SUMMARY:
The goal of this clinical trial is to learn about the effects of fluconazole in patients who plan to start or are currently undergoing standard of care treatment and plan to dose-escalate an IL-23 therapy for their Crohn's disease.

The main question it aims to assess is whether or not patient response to IL-23 therapies improve when simultaneously treated with fluconazole.

DETAILED DESCRIPTION:
The purpose of this study is to examine the efficacy and safety of fluconazole in combination with IL-23 therapy versus IL-23 therapy alone for the treatment of Crohn's disease (CD). IL-23 therapy may include ustekinumab (anti-interleukin-12/23), risankizumab (anti-interleukin-23), or guselkumab (anti-interleukin-23).

Subjects will be stratified into two groups based on standard of care treatment: IL-23 therapy initiation or IL-23 therapy dose escalation. Subjects in each group will then be randomized to one of two treatment arms:

1. IL-23 Therapy with Fluconazole (200 mg on Day 0 and 100 mg on Days 1-13)
2. IL-23 Therapy with Placebo (200 mg on Day 0 and 100 mg on Days 1-13)

Subjects will blindly receive the fluconazole treatment only if they meet all inclusion and exclusion criteria. Subjects will return for standard of care clinic visits 2 weeks post-treatment initiation and 12 weeks post-treatment initiation. Disease activity will be assessed at standard of care visits. Stool, blood, and oral swab samples will collected for research from subjects at Day 0 (pre-treatment initiation), Week 2 post-treatment initiation, Week 8 post-treatment initiation, and Week 12 post-treatment initiation. If subjects consent to biopsies, biopsies will also be collected for research at endoscopic procedures (colonoscopies and/or flexible sigmoidoscopies). Subjects will return at Week 24 and 1 year post-treatment initiation for standard of care visits, where blood, stool, and oral swabs will also be collected for research.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at least 18 years old
2. Patients with mild to moderate Crohn's disease as defined by CDAI score of 150-450

Exclusion Criteria:

1. Antifungal usage within one month prior to initiation of blinded fluconazole usage
2. Known allergy to fluconazole
3. Patients with known hepatic disease, cirrhosis, or with elevated liver biochemistries (e.g., transaminase(s) >3X upper limit of normal (ULN), and/or bilirubin levels >1.5X ULN (with exception of confirmed Gilbert's disease) at baseline
4. Patients taking any medications judged by clinical provider to interact with fluconazole and are known contraindications (refer to section 2.2) and cause serious adverse events, including but not limited to death, cardiac events, serious cardiac dysrhythmias, and prolongation of QTc
5. Pregnant or lactating women
6. Severe Crohn's disease defined by a PRO-2 score ≥ 34 or imminent need for surgery, or deemed not medically fit by physician
7. Patient with symptomatic stricturing
8. Patient with pouchitis or an ostomy
9. Patients with known, active fungal infection(s) since these patients would require particular, standard-of-care monitoring and treatment, which may include intravenous and/or prolonged courses of fluconazole or other therapies.
10. Patients with hypokalemia, or advanced cardiac failure
11. Patients with renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving clinical response | Week 12 post-Fluconazole Initiation
  Participants with clinical response are those participants with a reduction of the Crohn's Disease Activity Index (CDAI) by 100 or more points from baseline at week 12 post-Fluconazole initiation.

SECONDARY OUTCOMES:
Proportion of subjects achieving clinical remission | Week 12 post-Fluconazole Initiation
  Participants achieving clinical remission are those participants with a Crohn's Disease Activity Index (CDAI) score of no greater than 150 points at week 12 post-Fluconazole initiation.
Proportion of patients achieving endoscopic response or remission | Up to 1 Year post-Fluconazole Initiation
  Participants achieving endoscopic response are those participants with a reduction in the Simple Endoscopic Score for Crohn's Disease (SES-CD) of at least 50% from baseline. Participants achieving endoscopic remission are those participants with an SES-CD score less than or equal to 2

CONTACTS AND LOCATIONS:
Overall Officials: Randy Longman, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No